CLINICAL TRIAL: NCT01086670
Title: Physical, Functional and Neural Effects of Two Lower Extremity Exercise Programs in Children With Cerebral Palsy
Brief Title: Physical, Functional and Neural Effects of Two Lower Extremity Exercise Protocols in Children With Cerebral Palsy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100073; 10-CC-0073
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Cerebral Palsy; Children; Adolescents
Keywords: Coordination; Neuroimaging; Motion Analysis; Locomotor
MeSH Terms: conditions — Cerebral Palsy | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 1 (Other): Subjects will be randomly assigned to use one of two novel lower extremity exercise devices: a motor-assisted cycle or an elliptical trainer.
  Interventions: Other: Physical Exercise

INTERVENTIONS:
Other: Physical Exercise — Children will be assigned either an elliptical machine or cycle to take home. Each exercise will be performed for 20 minutes per day, 5 days per week for a period of 12 consecutive weeks, or 60 sessions in all. To avoid excessive fatigue or over-training effects, children are asked to adhere to this exact schedule and not to exercise more than this. Children are asked to complete as many of the sessions as they can. To allow for sick days or vacation during the program, the duration of the training can be extended up to 2 more weeks if needed to try to complete all 60 sessions. Compliance (percent sessions completed) will be correlated with outcomes in the statistical analyses.

SUMMARY:
Background:

* Many people who have cerebral palsy (CP) have spastic diplegia, which affects the legs and causes difficulty with leg movement and walking. Research has shown that exercise can help those with CP learn to move their arms better, but more research is needed to determine whether exercise programs can improve leg movements in people with CP.
* Walking on a treadmill with the help of a physical therapist has improved the treatment outcomes of some individuals with spinal cord injuries. Many children with CP already have physical therapy but still have trouble with walking and leg coordination. Two other kinds of exercise machines, a stationary bicycle and an elliptical machine, used in the home, may be able to help children with CP walk better and move their legs better.

Objectives:

* To see how children with cerebral palsy (CP) move their legs differently from children without CP.
* To see if an exercise program can improve leg coordination in children with CP.

Eligibility:

- Children between 5 and 17 years of age who either have spastic diplegia CP or are healthy volunteers.

Design:

* Children who are able and willing will have magnetic resonance imaging (MRI) scans at the start and the end of the study.
* During Part I of the study, participants will demonstrate their leg and muscle function with the following tests:
* Measurement of leg size and movement
* Combined camera motion study and electrical impulse evaluation to assess how well the participant walks (with or without an assistive device, as needed)
* Leg movement tests on an exercise bicycle and elliptical machine
* Tests of leg muscle strength, stiffness, and effectiveness
* Ultrasound scans of leg muscle
* Parents of participants will complete computer-based questionnaires about their child s motor abilities.
* A smaller group of participants will continue to Part II of the study, which involves regular exercise of 20 minutes a day, 5 days a week, for 3 months, on a stationary bicycle or elliptical trainer. Half of the group will start this exercise program immediately after the first part of the study, while the other half will wait 3 months before beginning the exercise program.
* During Part II, participants will return to the clinical center for two more sets of the tests and evaluations performed in Part I.

DETAILED DESCRIPTION:
Objectives:

Our primary objectives are to: 1) characterize and compare lower extremity motor coordination in children with cerebral palsy (CP) across mobility levels and to children without CP; and 2) evaluate the effects of two home-based exercise programs on motor coordination, as well as other physical, functional and neurological outcomes in children with CP. We hypothesize children with CP will exhibit significant coordination deficits compared to those without CP and that each exercise program will lead to significant improvements in outcomes.

Study Population:

Objective 1 will include 60 ambulatory children with spastic diplegic CP (20 in each of three mobility levels) and 20 children without CP within the same age range. Forty (40) children with CP will participate in Objective 2; 20 in each exercise group.

Design:

In Objective 1, the multiple measures taken at a single point in time will be compared across the three CP and the control groups. Children with CP from Objective 1 will be invited consecutively to participate in the exercise program (Objective 2), until enrollment is complete. Participation in Objective 2 lasts for 6 months. Subjects will be randomly assigned to use one of two novel lower extremity exercise devices: a motor-assisted cycle or an elliptical trainer. Children will exercise for 20 minutes, 5 days a week for 12 consecutive weeks. The major goal of each is to increase the ability to cycle or step at a rapid pace (the target goal is 40 RPM), with resistance added once speed goals are attained and thereafter progressed gradually. The timing of the exercise period (immediate vs. delayed for 3 months) will also be randomly assigned allowing assessors to be masked to group assignment.

Outcome Measures:

The primary outcome is the difference (Objective 1) or pre to post-exercise change (Objective 2) in coordination as measured by the fastest active (voluntary) cadence with each device. Additional coordination measures include cadence at free speed, variability in cadence, and EMG reciprocation vs. synchronization. Selective Control Assessment for the Lower extremity (SCALE), strength and spasticity tests and ultrasound measures of muscle size will be assessed at each time point. These will be compared across groups and before and after the two exercise programs. Functional outcomes include gait speed and two validated computer-based questionnaires. Neural outcomes include selected measures of gray and white matter connectivity as assessed with fcMRI and DTI, respectively.

ELIGIBILITY:
* INCLUSION CRITERIA:

A. For those without CP (healthy volunteers)

1. Must be between the ages of 5-17, inclusive
2. Must be in good general health
3. Must be able to understand and comply with the requirements of the study

B. For those with CP

1. Must be between the ages of 5-17, inclusive
2. Have a diagnosis of spastic bilateral cerebral palsy
3. Documentation on previous MRI of peri-ventricular white matter injury
4. Able to walk at least 20 feet without stopping and without the need for assistance by another person. A hand-held assistive device (e.g. cane, walker) may be used if necessary.
5. Be able to understand and comply with the requirements of the study
6. Availability of an adult who agrees to be primarily responsible for completing the reporting requirements for the study and supervising the exercise program

EXCLUSION CRITERIA:

A. For those without CP (healthy volunteers)

1. Have a history of musculoskeletal or neurological injury or disorder or general medical condition that would affect the use of the legs or limit the ability to safely perform motor testing

B. For those with CP:

1. Receiving oral or intrathecal baclofen, which may depress neural plasticity, at the time of enrollment or during the study period
2. Had surgery to the lower extremities in the past year or any major surgery within the past 6 months
3. Presence of any major medical illness that would limit the ability to safely tolerate the exercise program
4. Requiring or desiring to have botulinum toxin injections within four months before or at any time during the study period.
5. Requiring the use of a device that provides support of the pelvis when walking (e.g. gait trainer)
6. If choosing to participate in the exercise program, cannot be currently using an exercise machine or start using one during the study period.

ADDITIONAL EXCLUSION CRITERIA FOR THOSE HAVING A MRI:

1. Pregnancy: For any female of childbearing potential who is not pregnant, a pregnancy test will be done.
2. A ventriculo-peritoneal shunt
3. Claustrophobia
4. Metal fragments, wires or implants in the brain or in any part of the skin or body
5. Excessive startle reaction to or fear of loud noises
6. Inability to remain still and quiet for up to five minutes at a time
7. Inability to be off levodopa for at least 24 hours

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2010-03-30 (Actual); Primary Completion 2015-01-12 (Actual); Study Completion 2016-05-09 (Actual)

PRIMARY OUTCOMES:
Coordination as measured by fast cadence during device and walking | per test, 3 months post test, 3 months follow up
  Cadence is the number of device cycles or gait cycles performed in a minute.

SECONDARY OUTCOMES:
3D Motion Capture of walking, cycling and elliptical, Surface electromyography, Selective Control Assessment of Lower Extremities, Physical examination, Muscle Ultrasound. strength and spasticity, Questionnaires, Magnetic Resonance Imaging | 12 weeks
  Tests will be presented in the same order at each assessment, with the 3D motion assessments of the cycling and steppingperformed first since these involve collection of the primary outcome measure, cadence.

CONTACTS AND LOCATIONS:
Overall Officials: Diane L Damiano, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2010-CC-0073.html